CLINICAL TRIAL: NCT04581980
Title: Modulation of Ghrelin Release by Exercise Intensity: The Role of Obesity and Prediabetes Status
Brief Title: Effects of Obesity and Intensity of Exercise on Ghrelin Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Arthur L Weltman, Dr. Arthur Weltman, Professor of Kinesiology, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 200241; 5R01DK129510-02 (NIH)
Record Dates: First submitted 2020-10-01; First posted 2020-10-09 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Insulin Resistance; Cardiovascular Risk Factor
Keywords: exercise; ghrelin; insulin resistance; vascular function; obesity; prediabetes
MeSH Terms: conditions — Obesity; Insulin Resistance; Motor Activity; Prediabetic State | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized, crossover design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): This arm will receive no exercise
- Moderate Intensity Exercise (Experimental): This group will exercise on a cycle ergometer (Lode Bike) at moderate intensity. Moderate intensity will be defined by the lactate threshold. A heart rate monitor will be utilized at all times to record heart rate.
  Interventions: Other: Exercise
- High Intensity Exercise (Experimental): This group will exercise on a cycle ergometer (Lode Bike) at high intensity. High intensity will be defined by an by 75% of the difference between the lactate threshold and peak.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants will exercise on a cycle ergometer
  Arms: High Intensity Exercise; Moderate Intensity Exercise

SUMMARY:
This study is investigating the effect of different intensities of exercise on levels of the hormone, ghrelin. In addition, we will be examining the relationship between any exercise induced changes in ghrelin and insulin sensitivity, obesity, and vascular function.

DETAILED DESCRIPTION:
The goal of this proposal is to characterize the effects of two exercise "intensity doses" on total ghrelin, acyl ghrelin, and des-acyl ghrelin in lean and obese adults with and without prediabetes. Ghrelin (TG) is involved in the regulation of appetite, energy balance, glucose metabolism and insulin sensitivity. Ghrelin exists in the blood in a des-acyl form (DAG ~78% of TG), and in an acylated form (AG ~22% of TG). Despite being less abundant, AG is has multiple actions that promote energy storage, including stimulation of appetite, inhibition of insulin release from the pancreas, and increases in adiposity via a widely characterized growth hormone secretagogue receptor. Conversely, DAG often opposes AG promoting negative energy balance (appetite suppression and reduced fat mass (FM)) and improving insulin sensitivity, acting through a receptor not yet identified. The optimal ratios of TG, DAG, and AG are not clear. Likewise, there is a need for targeted approaches that can effectively manipulate these peptides to aid in the prevention and/or treatment of obesity, metabolic syndrome, prediabetes and type 2 diabetes. Exercise provides a unique therapeutic approach in the treatment of dysregulated ghrelin.

Limited animal and human studies examining exercise and ghrelin release are mostly equivocal or only document TG and/or a single (e.g. AG) form of ghrelin. As DAG and AG can act synergistically, antagonistically, or have independent effects, the quantification of these peptides in response to exercise is critical to understanding the role of exercise on ghrelin release and ghrelin's exercise induced influence on overall glucose regulation and energy balance. Exercise intensity may be key, as exercise that elevates levels of lactate suppress AG and appetite post exercise. Here we propose to address this gap in knowledge by defining the role of acute exercise intensity, at doses above and below the lactate threshold, on TG, AG, and DAG release in lean and obese individuals with and without prediabetes. Specific Aim 1: Examine effects of exercise intensity on ghrelin, insulin, glucose and self-reported appetite. Hypothesis: Higher exercise intensity will result in differential effects on TG, AG, DAG, AG/DAG, insulin, and glucose AUC's, and appetite; affected by sex, obesity, abdominal visceral fat (AVF), and prediabetes status. Specific Aim 2: This is an exploratory aim using regression modeling to examine exercise-induced changes in ghrelin on glucose, insulin and appetite. Hypothesis: TG, AG, DAG and AG/DAG alterations will differentially predict changes in glucose metabolism, insulin sensitivity, and appetite. These alterations vary by sex, levels of obesity, AVF, and prediabetes. Results from this pilot/feasibility application will inform a larger submission that defines therapeutic exercise targets for TG, AG, and DAG, and examines the effects of individualized exercise training using precision exercise prescription techniques on ghrelin release.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* BMI between 18-40 kg/m2
* Untrained (reports less than 2 days/week of exercise)
* Weight stable (no significant loss/gain of more than 3kg in the past 3 months)
* Females must be premenopausal and report normal menstrual cycles

Exclusion Criteria:

* History of diabetes, gastrointestinal disease, or endocrine disorder
* Smoking (must have quit at least 6 months prior)
* Disordered eating
* Females currently pregnant or undergoing fertility treatments
* The following medications (due to their effect on insulin sensitivity ,endothelial function and/or ghrelin secretion): Synthetic growth hormone, metformin, synthetic insulin, sulfonylureas, meglitinides, Thiazolidinediones, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors , biguanides, alpha-glucosidase inhibitors, phosphodiesterase inhibitors, beta-blockers, alpha-blockers, ACE-inhibitors, ARB's, fibrates, glucocorticoids, olanzapine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Ghrelin | Measured at 6 timepoints over 2-3 hours during each experimental visit
  We will be analyzing plasma levels of acylated and deacylated ghrelin

SECONDARY OUTCOMES:
Appetite Questionnaire (VAS) | Measured at 6 timepoints over 2-3 hours during each experimental visit
  We will see how appetite may or may not change in response to exercise
Vascular Function (brachial flow mediated dilation) | Measured at 5 timepoints over 2-3 hours during each experimental visit
  We will be measuring how the arteries respond (i.e. dilate) in response to exercise

OTHER OUTCOMES:
Insulin Sensitivity | Insulin and glucose will be collected at 5 timepoints during the OGTT, and 11 timepoints during each testing visit. The Matsuda index (mathematical model) will be used to calculate insulin sensitivity
  We want to create a linear regression model to explore the relationship between exercise induced changes in ghrelin and insulin sensitivity
Body Composition | Body composition will be measured twice during a DEXA and CT scan (takes about 30 minutes)
  We want to create a linear regression model to explore the relationship between exercise induced changes in ghrelin and body composition (i.e. fat mass)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No